CLINICAL TRIAL: NCT01990027
Title: Swiss Kidney Stone Cohort (SKSC)
Acronym: SKSC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Swiss National Centre of Competence in Research Kidney Control of Homeostasis (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-2013-0330
Record Dates: First submitted 2013-10-09; First posted 2013-11-21 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Kidney Stone
Keywords: kidney stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Whole blood; plasma; serum; urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SKSC Patients group: A group a 1000 subjects affected by kidney stone as described in the eligibility criteria will be recruited in the period 2014-2024 and the same exams will be repeated for each participants for a period of 3 years.
  No intervention will be undertaken.
- SKSC Control group: A group of 250 stone-free participants will be recruited and analysed with the same protocol as the patients but in a single visit. This group will be used for comparison with the patients group in future studies.
  No intervention will be undertaken.

SUMMARY:
The SKSC is a continuous database with the objective of a standardized diagnosis and monitoring of patients with kidney stones as well as the establishment of a Biobank.

DETAILED DESCRIPTION:
The objective of this study is multi-site, standardized observation and characterization of kidney stone patients.

Furthermore, an adequate structure should be established for the execution of studies with kidney stone patients, in order to then, if necessary, develop recommendations for useful monitoring or prophylactic measures, as well as new treatment options for kidney stone patients.

A control group of 250 stone-free volunteers matching patients cohort participants for sex and age started recruitment in October 2017 and will serve the purpose of comparison in future studies.

ELIGIBILITY:
For SKSC Patients Group:

Inclusion Criteria:

Only patients that meet all of the following inclusion criteria can be included in this study:

* Signed Declaration of informed consent
* Male or female
* Recurrent kidney stone episodes (more than 1) or an individual kidney stone episode with one or several of the following risk factors:
* The first manifestation at the a minimum age of 25
* Positive family history
* Non-calcium oxalate stones
* Gastrointestinal disorders (e.g. gastric bypass surgery, inflammatory bowel disease, malabsorption etc.)
* Osteoporosis
* Nephrocalcinosis
* Single kidneyness
* Currently pregnant
* Gout
* Metabolic syndrome ( Diabetes Mellitus type I and II )
* Residual calculi (at least 3 months after the therapy)
* Bilateral or multiple stones
* Chronic urinary tract infection
* Chronic renal failure (eGFR lower than 60 ml/min.)
* Kidney transplant

Exclusion Criteria:

Patients with at least one of the following exclusion criteria may not take part in this study.

* Not signed Informed Consent form
* Age below 18 years old

For SKSC Control Group

Inclusion criteria:

* Signed Declaration of informed consent
* Male or female
* Kidney-stone free (screening verification by low-dose CT-scan)

Exclusion criteria:

* Not signed Informed Consent form
* Age below 18 years old
* Pregnancy
* History of kidney stones
* Low-dose CT-scan positive for kidney stones during screening phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a kidney stone episode + Kidney stone-free control group
Sampling Method: Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2014-04; Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Epidemiological characterization | 10 years
  Epidemiological characterization of kidney stone patients

CONTACTS AND LOCATIONS:
Locations (6):
- Switzerland (6):
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - HUG, Geneva, Canton of Geneva
  - USZ, Zurich, Canton of Zurich
  - Universitätsspital Basel, Basel
  - Inselspital, Bern
  - CHUV, Lausanne

REFERENCES:
- [Derived] Roth B, Bonny O; Swiss Kidney Stone Cohort Investigators. The Swiss Kidney Stone Cohort: An Observational Study to Unravel the Cause of Renal Stone Formation. Eur Urol Focus. 2017 Feb;3(1):7-9. doi: 10.1016/j.euf.2017.03.003. Epub 2017 Mar 21. PMID 28720370
- See also: Related Info — http://nccr-kidney.ch